CLINICAL TRIAL: NCT06453733
Title: Crainio Non-invasive Intracranial Pressure Monitor for Traumatic Brain Injury: Product Development
Brief Title: Crainio Non-invasive ICP Monitor for TBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Crainio Ltda (Industry)
Collaborators: Innovate UK (Other Government); Barts & The London NHS Trust (Other); City, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 341050
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Traumatic Brain Injury
Keywords: Intracranial pressure; Non-invasive monitoring; Machine learning; Photoplethysmography
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crainio (Experimental): Acquisition of cerebral PPG signals from Crainio's probe stuck to the patient's forehead, alongside concurrent invasive ICP measurements in patients with traumatic brain injury
  Interventions: Device: Crainio

INTERVENTIONS:
Device: Crainio — Crainio device comprises a forehead-mounted sensor containing infrared light sources that can illuminate the deep brain tissue of the frontal lobe. Photodetectors in the sensor detect the backscattered light, which is modulated by pulsation of the cerebral arteries. A control unit processes the backscattered light (called the photoplethysmogram, PPG) and transmits it to a computer device to train ML models that will estimate ICP offline.
  Other Names: nICP probe, Crainio system

SUMMARY:
The clinical investigation aims to advance the Crainio device, designed for non-invasive intracranial pressure (ICP) monitoring. This feasibility study involves 54 participants over a 12-month period and seeks to collect cerebral photoplethysmogram signals alongside concurrent invasive ICP measurements in patients with traumatic brain injury. The primary objective is to establish the diagnostic accuracy of the Crainio device, aiming for at least 90% sensitivity and specificity in detecting raised ICP (above 20 mmHg). Secondary objectives include evaluating patient-related factors such as skin tone, skull thickness, and skull density, as well as the tolerability and acceptance of the device by both patients and healthcare professionals.

DETAILED DESCRIPTION:
Intracranial pressure (ICP) is routinely monitored in patients suffering from traumatic brain injury (TBI). Raised ICP can result in compression of the cerebral vasculature and subsequent reduction in oxygen and nutrient delivery to the brain leading to significant morbidity and mortality. In fact, raised ICP is the most common cause of death in patients with severe TBI.

Standard ICP monitoring requires insertion of a cranial bolt into the skull through which an electrical transducer is inserted. Alternatively, an intra-ventricular catheter is inserted through a burr hole. Both of these monitoring methods are associated with risks including haemorrhage and infection, as well as delay in establishing emergency monitoring and limiting it to hospitals that have neurosurgery.

There has been much research in recent years to find a method for measuring intracranial pressure noninvasively (nICP), including measurement of pressure in the retinal veins, measurement of eardrum displacement, transcranial Doppler ultrasonography and imaging-based solutions. These methods all require considerable user intervention and are non-continuous.

This project aims to collect cerebral photoplethysmogram signals and concurrent invasive ICP measurements from patients with traumatic brain injury to develop Crainio machine learning (ML) algorithms. The core intellectual property (IP) of this continuous external monitoring ICP system was originally developed by academics in the lab of Professor Kyriacou at City, University of London. Crainio is a spin-out company that was created to industrialise and commercialise this research on an exclusive basis.

The device comprises a forehead-mounted sensor containing infrared light sources that can illuminate the deep brain tissue of the frontal lobe. Photodetectors in the sensor detect the backscattered light, which is modulated by pulsation of the cerebral arteries. A control unit processes the backscattered light (called the photoplethysmogram, PPG) and transmits it to a computer device to train ML models that estimate an absolute value of ICP.

The basic science behind this method for measuring ICP is that changes in the extramural arterial pressure affect the morphology of the recorded optical pulse, so analysis of the acquired signal using an appropriate algorithm will enable calculation of nICP. The reported nICP will provide screening at the triage stage, indicating the need for imaging or rapid intervention (such as haematoma evacuation) and guide head injury management, notably ICP-targeted treatment regimes. Ultimately this could lead to significant improvements in secondary injury-related mortality, length of hospital stay and reduced post-trauma disability.

This feasibility study aims to collect the clinical data with which to train the nICP algorithms to the point that they can detect raised intracranial pressure (ICP>20 mmHg) with sufficient sensitivity and specificity that Crainio device can be regulated for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of traumatic brain injury.
* Adults (aged between 16 and 99, male and female)
* TBI patients admitted to the Royal London Hospital.
* Patients having invasive ICP monitoring as part of their normal medical treatment.

Exclusion Criteria:

* Forehead skin is not intact.
* Decompressive craniectomy patients.
* Open external ventricular drainage (EVD) treatment.
* Patients who will unlikely survive the following twelve hours.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 12 hours record per patient
  Generate a nICP model offline with a sensitivity above 90% to discriminate ICP values over 20 mmHg.
Specificity | 12 hours record per patient
  Generate a nICP model offline with a specificity above 90% to discriminateICP values over 20 mmHg.

SECONDARY OUTCOMES:
Skin tone through Fitzpatrick scale | 1 classification per patient (3 minutes)
  Evaluating the effect on the nICP model of patient-related factors such as the skin tone.
Skull thickness through CT scan | 1 measurement per patient (3 minutes)
  Evaluating the effect on the nICP model of patient-related factors such as the skull thickness.
Skull density through Age stratification analysis | 1 classification per patient (1 minute)
  Evaluating the effect on the nICP model of patient-related factors such as the skull density.
Device usability | 1 form per patient (5 minutes)
  Customised form to assess the acceptance of the device by the healthcare proffesionals.
Advers effects and events | 12 hours record per patient
  Evaluate the device safety by monitoring the development of possible advers effects or events in the patients while data is acquired

CONTACTS AND LOCATIONS:
Overall Officials: Chris Uff, Dr, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Royal London Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the final results of Crainio device diagnostic accuracy and safety would be published. Any individual participant data would be available to other researchers.

REFERENCES:
- [Background] Roldan M, Kyriacou PA. Near-Infrared Spectroscopy (NIRS) in Traumatic Brain Injury (TBI). Sensors (Basel). 2021 Feb 24;21(5):1586. doi: 10.3390/s21051586. PMID 33668311
- [Background] Roldan M, Abay TY, Kyriacou PA. Non-Invasive Techniques for Multimodal Monitoring in Traumatic Brain Injury: Systematic Review and Meta-Analysis. J Neurotrauma. 2020 Dec 1;37(23):2445-2453. doi: 10.1089/neu.2020.7266. Epub 2020 Sep 24. PMID 32821023
- [Background] Roldan M, Chatterjee S, Kyriacou PA. Brain Light-Tissue Interaction Modelling: Towards a non-invasive sensor for Traumatic Brain Injury. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:1292-1296. doi: 10.1109/EMBC46164.2021.9630909. PMID 34891522
- [Background] Roldan M, Kyriacou PA. Head Phantom Optical Properties Validation for Near-Infrared Measurements: A Comparison with Animal Tissue. Annu Int Conf IEEE Eng Med Biol Soc. 2022 Jul;2022:641-644. doi: 10.1109/EMBC48229.2022.9871103. PMID 36085774
- [Background] Roldan M, Bradley GRE, Mejia-Mejia E, Abay TY, Kyriacou PA. Non-invasive monitoring of intracranial pressure changes: healthy volunteers study. Front Physiol. 2023 Aug 8;14:1208010. doi: 10.3389/fphys.2023.1208010. eCollection 2023. PMID 37614754
- [Background] Roldan M, Abay TY, Uff C, Kyriacou PA. A pilot clinical study to estimate intracranial pressure utilising cerebral photoplethysmograms in traumatic brain injury patients. Acta Neurochir (Wien). 2024 Feb 27;166(1):109. doi: 10.1007/s00701-024-06002-4. PMID 38409283
- [Background] M. Roldan and P. A. Kyriacou, Head Phantom for the Acquisition of Pulsatile Optical Signals for Traumatic Brain Injury Monitoring, Photonics, vol. 10, no. 5, 2023
- [Background] T. Y. Abay, J. P. Phillips, C. Uff, M. Roldan, and P. A. Kyriacou, In Vitro Evaluation of a Non-Invasive Photoplethysmography Based Intracranial Pressure Sensor, Appl. Sci., vol. 13, no. 1, p. 534, Dec. 2022
- [Background] M. Roldan and P. A. Kyriacou, "A non-Invasive Optical Multimodal Photoplethysmography-Near Infrared Spectroscopy Sensor for Measuring Intracranial Pressure and Cerebral Oxygenation in Traumatic Brain Injury," Appl. Sci., 2023